

## WRITTEN INFORMED CONSENT

Title of the study: Social Return on Investment Project (SROI) of the waiting list management system for surgery and diagnostic tests.

| have read and understood the information sheet given to me. |
|---|
| have been able to ask questions about the study. |
| I understand that my participation is voluntary. |
| I understand that I can withdraw from the study: |
| 3º Without this having any repercussions on my medical care. |
| I freely give my agreement to participate in the study. |



## **ORAL CONSENT IN FRONT OF WITNESSES**

| Title of the study: | Social | Return ( | on | Investment | Project | (SROI) | of | the | surgical | waiting | list | and |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| diagnostic tests management system. | | | | | | | | | | | | |
| I (name and surnam | e) | | | | | | | | | | | |

declare under my\_\_\_\_\_\_ responsibility that (name of participant in the study)

I have received the information sheet about the study.

I have been able to ask questions about the study.

I have received sufficient information about the study.

Has been informed by: José Luis González Muñoz.

You understand that your participation is voluntary.

You understand that you can withdraw from the study:

1º Whenever you want

2º Without having to give explanations.

3º Without this having any repercussions on your medical care.

And he/she has freely expressed his/her agreement to participate in the study.

| DATE: | |
|-------|--------------------------|
| | SIGNATURE OF THE WITNESS |



## **CONSENT OF THE REPRESENTATIVE**

| Titl | e of the | study: | Social Returr | n on Investment | t Project (SROI) of | the surgi | cal v | vaitin | g list and |
|---|---|---|---|---|---|---|---|---|---|
| dia | gnostic te | sts man | agement syst | tem. | | | | | |
| I | (name | and | surname) | | | ir | ١ . | the | capacity |
| of_ | | | (re | elationship to pa | rticipant) of | | | | |
| (na | me of stud | dy parti | cipant). | | | | | | |
| I ha | ave read a | nd unde | erstood the st | tudy information | sheet. | | | | |
| ۱w | as able to | ask que | stions about | the study. | | | | | |
| l re | ceived sat | isfactor | ry answers to | my questions. | | | | | |
| I ha | ave receive | ed suffic | cient informa | tion about the st | tudy. | | | | |
| I ha | ave spoker | n to: Jos | é Luis Gonzál | lez Muñoz. | | | | | |
| l ur | nderstand | that pa | rticipation is | voluntary. | | | | | |
| l ur | nderstand | that I ca | an withdraw f | from the study: | | | | | |
| 1º ' | Whenever | you wa | ant | | | | | | |
| 2º | Without h | aving to | give explana | ations. | | | | | |
| 3º ' | Without th | nis havii | ng any reperc | cussions on your | medical care. | | | | |
| In | my preser | nce, | | | _ (name of study p | participant) | has | been | n given all |
| rele | evant info | rmation | adapted to h | nis/her level of u | nderstanding and a | grees to pa | rtici | pate. | |
| An | d I agree | to | | | | _ (name o | f stu | dy pa | articipant) |
| par | ticipating | in this s | study. | | | | | | |
| D | ATE: | | | | | | | | |
| | | | SIC | GNATURE OF TH | E REPRESENTATIVE | | | | |